CLINICAL TRIAL: NCT00663988
Title: Human Partial Facial Allotransplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Guo Shuzhong, Xijing Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJ-GuoSZ0709
Record Dates: First submitted 2008-04-20; First posted 2008-04-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2006-02

CONDITIONS: Pharmaceutical Preparations
Keywords: face transplantation
MeSH Terms: interventions — TSTA3 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- III (Experimental): The effect of human partial facial allotransplantation
  Interventions: Procedure: human transplantation

INTERVENTIONS:
Procedure: human transplantation — Allograft composite tissue transplantation. procedure. medication
  Other Names: face allograft

SUMMARY:
Progress in composite tissue allotransplantation provides a new remedy for severely disfigured patients. We plan to carry out allograft composite tissue transplantation after a careful systemic preparation.

DETAILED DESCRIPTION:
Severe facial deformities caused by burn, trauma, or tumor resection, are usually organs defects, such as ear, nose, eyelid, or lips and tissue defects involving the skin, fat tissue, muscle, cartilage, or bone etc. The optimal reconstruction of these specialized units is difficult to achieve.1 The face is not simply a mask but a functional, dynamic and important aesthetic organ. The functions of face include talking, smiling, eating, and winking. The reconstructive challenge is complicated by the fact that the human eye looks for and can detect the slightest abnormality in another's face. Traditional reconstructive procedures include free skin graft, application of local flaps, tissue prefabrication, tissue expansion, and free tissue transfer. Despite the application of meticulous techniques and artistic creativity, even the most skillful surgeon cannot reproduce this most complex part of the body. Facial reconstruction is still a tough challenge to surgeons.

In recent years, with the progress in composite tissue allotransplantation, there comes a new hope for the severely disfigured patients. The apparent success in human hand allotransplantation in the late 1990s laid the immunological and ethical groundwork for performing human facial allotransplantation and let surgeons consider the use of donor facial tissues for reconstructing severe facial deformities.The outcome of hand and forearm transplantation has been more successful than might have been predicted but nevertheless there has been a quite high incidence of rejection, in general controlled by additional immunosuppression, and there has also been chronic rejection seen in some of cases5. But facial transplantation, which will inevitably encounter many problems, is different from hand transplantation. Reports of the Royal College of Surgeons of England outlined the problems and potential down side of face transplantation, which including technical failure, acute rejection, chronic rejection, side effects of immunosuppressive therapy, noncompliance with immunosuppressive medication, psychologic and societal issues, ethical issues, et al.So Jean-Michel Dubernard said that face transplantation was much more difficult than the hand technically.

To solve these problems, many experts conducted related studies. Ulusal et al built the first facial/scalp flap transplantation model of rat. Cyclosporine A was used to prevent acute and chronic allograft rejections after the transplantation. Experts used animal facial transplantation models to study blood supply, tolerance induction, donor-specific chimerism, and medication. Cleveland Clinic Foundation carried out a series of studies on cadaver for facial allograft transplantation in preparation for facial transplantation in humans.Since 2002, we have been studying facial transplantation and have built a half facial transplantation model in rabbit . We chose Ciclosporin A, Azathioprine and Prednisone as immunosupressants and got a good result. Since the late 1990s, the progresses of these studies have strongly suggested that facial transplantation is bound to success.

In November 2005, the first partial facial transplantation was carried out successfully and got a good result in Amiens, France.

The recipient, a 30 years old man, came from a remote village of Yunnan province, China. His face was scratched by a bear in October 2004. Shortly after the disaster, he was treated by debridement and repaired with left forearm pedicle flap. But efficacy of these conventional techniques was not satisfactory and facial wounds did not heal, which seriously affected his appearance and function, and even his normal work and life. He was arranged to stay in hospital for further examinations and treatments on March 11, 2006.

The major defections on the patient's face involved extensive skin and soft tissue in the right buccal division combined with severe cicatricial contracture deformity, upper lip, total nose, the front wall of the right maxillary sinus, the lateral right orbital wall and infraorbital wall, the right zygomatic bone, a large portion of the right parotid gland.

Examinations showed panel reaction antibody (PRA) was very high (99% and 98% in two separate examinations), which implied the recipient belonged to the highly sensitive crowd. It is well known that highly sensitive patients with PRA often present with acute rejections. To decrease PRA and also the risk of surgery, immunoadsorption column of Protein A was used. Reexaminations showed that PRA was below 5% (in two separate examinations) before the surgery. Other medical examinations showed there were no surgical contraindications.

For this patient, traditional reconstructive procedures, including free skin graft, application of local flaps, tissue prefabrication, tissue expansion, and free tissue transfer, can only cover the wound. Without bony framework, reconstruction of the nose is too hard by traditional procedures. And the reconstruction of the upper lip is hard too. Face transplantation can be an appropriate operative indication for this patient..

ELIGIBILITY:
Inclusion Criteria:

* normal function of heart/liver/kidney

  * donor: same boold type
  * at least 3 sites were matched within 6 HLA sites

Exclusion Criteria:

* abnormal function of heart/liver/kidney

  * donor: not the same boold type and 1 or 2 sites were matched within 6 HLA sites

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2006-04; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
improved health | 1 M

SECONDARY OUTCOMES:
improvement of abnormal states | 3 Y

CONTACTS AND LOCATIONS:
Overall Officials: Shuzhong Guo, Dr, Study Director — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Dubernard JM, Lengele B, Morelon E, Testelin S, Badet L, Moure C, Beziat JL, Dakpe S, Kanitakis J, D'Hauthuille C, El Jaafari A, Petruzzo P, Lefrancois N, Taha F, Sirigu A, Di Marco G, Carmi E, Bachmann D, Cremades S, Giraux P, Burloux G, Hequet O, Parquet N, Frances C, Michallet M, Martin X, Devauchelle B. Outcomes 18 months after the first human partial face transplantation. N Engl J Med. 2007 Dec 13;357(24):2451-60. doi: 10.1056/NEJMoa072828. PMID 18077810
- [Result] Xudong Z, Shuzhong G, Yan H, Datai W, Yunzhi N, Linxi Z. A hemifacial transplantation model in rabbits. Ann Plast Surg. 2006 Jun;56(6):665-9. doi: 10.1097/01.sap.0000202829.24619.19. No abstract available. PMID 16721082